CLINICAL TRIAL: NCT00373724
Title: A Placebo-Controlled Study Assessing Lateral Branch Radiofrequency Denervation for Sacroiliac (SI) Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 05-03-23-05
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Low Back Pain
Keywords: sacroiliac joint; low back pain; radiofrequency
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: radiofrequency denervation

SUMMARY:
In order to determine whether L4 and L5 primary dorsal rami and S1-3 lateral branch radiofrequency denervation is effective for sacroiliac (SI) joint pain, we are conducting a randomized, controlled study.

DETAILED DESCRIPTION:
30 subjects with SI joint pain confirmed by SI joint injections will be randomized to receive either L4 and L5 primary dorsal rami and S1-3 lateral branch radiofrequency denervation or sham denervation. To facilitate patient blinding, in both groups 1 ml of lidocaine will be injected before true (or sham) denervation so patients cannot feel heating. The stimulation will be the same for both groups and blinding assessed after the procedure. Follow-up visits will be at 1,3 and 6-months postprocedure.

ELIGIBILITY:
Inclusion Criteria:

* Sacroiliac joint pain
* Age > 18

Exclusion Criteria:

* No focal neurological signs or symptoms, coagulopathy, unstable medical or psychiatric condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-11; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
visual analogue scale pain score, Oswestry Disability Index | 1, 3 and 6 months postprocedure

SECONDARY OUTCOMES:
Medication reduction, global perceived effect, work status

CONTACTS AND LOCATIONS:
Overall Officials: Steven P Cohen, MD, Principal Investigator — Johns Hopkins School of Medicine; Srinivasa N Raja, MD, Study Director — Johns Hopkins School of Medicine
Locations (2):
- United States (2):
  - Walter Reed Army Medical Center, Washington D.C., District of Columbia
  - Johns Hopkins School of Medicine, Baltimore, Maryland

REFERENCES:
- [Background] Cohen SP, Abdi S. Lateral branch blocks as a treatment for sacroiliac joint pain: A pilot study. Reg Anesth Pain Med. 2003 Mar-Apr;28(2):113-9. doi: 10.1053/rapm.2003.50029. PMID 12677621
- [Background] Yin W, Willard F, Carreiro J, Dreyfuss P. Sensory stimulation-guided sacroiliac joint radiofrequency neurotomy: technique based on neuroanatomy of the dorsal sacral plexus. Spine (Phila Pa 1976). 2003 Oct 15;28(20):2419-25. doi: 10.1097/01.BRS.0000085360.03758.C3. PMID 14560094
- [Background] Cohen SP. Sacroiliac joint pain: a comprehensive review of anatomy, diagnosis, and treatment. Anesth Analg. 2005 Nov;101(5):1440-1453. doi: 10.1213/01.ANE.0000180831.60169.EA. PMID 16244008
- [Derived] Cohen SP, Hurley RW, Buckenmaier CC 3rd, Kurihara C, Morlando B, Dragovich A. Randomized placebo-controlled study evaluating lateral branch radiofrequency denervation for sacroiliac joint pain. Anesthesiology. 2008 Aug;109(2):279-88. doi: 10.1097/ALN.0b013e31817f4c7c. PMID 18648237